CLINICAL TRIAL: NCT03037749
Title: Over-arousal as a Mechanism Between Alcohol and Intimate Partner Violence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Brandi C. Fink, PhD, Assistant Professor, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-433
Record Dates: First submitted 2016-04-19; First posted 2017-01-31 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Domestic Violence; Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: This is a within subjects design where distressed violent and distressed nonviolent partners participated in a placebo-controlled alcohol administration study with an emotion-regulation task.
Who Masked: Participant
Masking Description: Both distressed violent and distressed nonviolent partners participated in two experimental sessions and were counter-balanced to receive either an alcohol beverage or a placebo beverage in the first or second experimental session.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distressed violent (Experimental): Distressed violent partners participated in a within-subjects placebo-controlled alcohol administration arm with an emotion-regulation task.
  Interventions: Drug: Alcohol beverage; Drug: Placebo beverage
- Distressed nonviolent (Experimental): Distressed nonviolent partners participated in a within-subjects placebo-controlled alcohol administration arm with an emotion-regulation task.
  Interventions: Drug: Alcohol beverage; Drug: Placebo beverage

INTERVENTIONS:
Drug: Alcohol beverage — Alcohol beverage measured to have participant achieve a BAC of 0.08%
Drug: Placebo beverage — Placebo beverage measured to mimic the smell and taste of the alcohol beverage.

SUMMARY:
Intimate partner violence (IPV) is a serious public health problem costing $8.3 billion per year with over $6 billion in direct medical and mental health costs alone. Alcohol is present in most incidents of IPV, and contributes to more frequent and severe IPV incidents. These facts, coupled with the fact that there are no effective interventions for IPV, make understanding mechanisms through which alcohol is associated with IPV critical.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a significant public health problem for which there are currently no effective treatments. Alcohol use is present in most instances of IPV and is associated with an increase in the frequency and severity of IPV. The investigators believe that alcohol may be related to the increase in frequency and severity of IPV through a process of over-arousal that results from the cortically and psychophysiological arousing effects of alcohol during the ascending limb of intoxication and at peak Blood Alcohol Concentration (BAC) compounded by the unique behavioral and affective patterns of violent couples. The first aim of the proposal is to determine if increases in arousal after alcohol exposure is potentiated by evocative partner stimuli and is greater for distressed violent (DV) partners than distressed nonviolent (DNV) partners. A second aim is to determine if alcohol induced arousal interferes with DV partners' ability to regulate emotion in response to evocative partner stimuli compared to DNV partners. The proposed study is an experimental comparison of the effects of alcohol on arousal and emotion regulation between 35 DV and 35 DNV partners. One partner from each DV couple will be pseudo-randomly selected and yoked to a DNV partner of the same sex and comparable relationship satisfaction for participant in the experiment. To test the overall hypothesis that over-arousal is a mechanism through which alcohol is associated with increases in the frequency and severity of IPV, the selected partners will participate in a counter-balanced placebo session and an alcohol administration session during which electroencephalography (EEG), psychophysiology and pupillary response measurements of arousal will be collected during an emotion regulation task. The data will be analyzed using a repeated measures ANOVA with a between-subjects factor. The investigators expect that DV partners will experience significantly greater arousal than DNV partners during the evocative stimuli condition. The investigators also expect that DV partners will experience greater difficulty regulating emotion during evocative stimuli than DNV partners and that this effect will be compounded during the alcohol administration condition. Findings from this study will provide firm evidence that alcohol is associated with IPV through a mechanism of over-arousal and provide key targets for intervention to prevent future IPV. The data from the current proposal will be used to test biofeedback as an adjunct to a novel behavioral intervention to reduce drinking and increase behavioral flexibility in couples with a history of IPV.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Heterosexual,
* Be in a distressed relationship
* consume at least one to two alcoholic drinks per sitting each week for females and three to four alcoholic drinks for males
* report two binge drinking episodes (>4 drinks for males, >3 drinks for females) in month prior to assessment
* be married or cohabitating for at least six months
* both partners must be willing to participate
* must have a breath alcohol level of 0.0 g% at all visits.
* Distressed Violent couples must have a history of at least mild physical aggression in the past six months (e.g.,twisted partner's arm or hair).

Exclusion Criteria:

* currently separated
* an order of protection in place
* facing violence-related criminal charges
* currently in a domestic violence shelter
* evidence of psychosis or severe personality disturbance
* pregnant
* taking a medication contraindicated for use with alcohol
* currently taking insulin or oral hypoglycemic medication,
* an AUDIT score greater than 19 indicating dependent drinking
* illicit drug use (except marijuana)
* provide a positive urinalysis at first emotion-regulation session

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09-27 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
neurophysiological arousal collected via electroencephalography | two years
  electroencephalography. Each participant's individual neurophysiological responses will be collected and then aggregated at the conclusion of the study for between-group analyses. Greater alpha and beta frequencies relative to reduced to theta and delta frequencies indicate greater cortical arousal. The experimental conditions of this study will allow us to determine if distressed violent partners experience greater cortical arousal in certain conditions.
neurophysiological arousal collected via electrocardiogram | two years
  respiratory sinus arrythymia. This is a measure of heart rate variability that is an index of a person's ability to regulate their emotion. The responses on this measure are evaluated against the comparison group. Each participant's individual neurophysiological responses will be collected and then aggregated at the conclusion of the study for between-group analyses.
neurophysiological arousal collected via galvanic skin response | two years
  galvanic skin response. When people are neurophysiologically aroused, their skin sweats more. This responses on this measures these changes between conditions and groups, and are evaluated against the comparison group. Each participant's individual neurophysiological responses will be collected and then aggregated at the conclusion of the study for between-group analyses.
neurophysiological response collected via respiration | two years
  respiration. When neurophysiologically aroused people breathe faster. This responses on this measure will are evaluated against the comparison group to determine if the distressed violent group is more neurophysiologically aroused in certain experimental conditions. Each participant's individual neurophysiological responses will be collected and then aggregated at the conclusion of the study for between-group analyses.
neurophysiological response collected via eye tracking | two years
  pupillary response. When people are neurophysiologically aroused their pupils dilate. This responses on this measure are evaluated against the comparison group. Each participant's individual neurophysiological responses will be collected and then aggregated at the conclusion of the study for between-group analyses.
emotion regulation | two years
  This is an experimental task that all participants in both the distressed violent group and the distressed nonviolent group complete. In the emotion regulation task, an comparison of the aggregated primary outcome measures will be compared between groups to determine if distressed violent participants experience greater neurophysiological arousal than distressed nonviolent participants.

CONTACTS AND LOCATIONS:
Overall Officials: Brandi C Fink, Ph.D., Principal Investigator — University of Oklahoma; Eric D. Claus, Ph.D., Principal Investigator — The Mind Research Network
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03037749/Prot_SAP_ICF_000.pdf